CLINICAL TRIAL: NCT02721992
Title: A Prospective Study on the Association Between Graves' Orbitopathy and Hypercholesterolemia
Brief Title: Graves' Orbitopathy and Hypercholesterolemia
Acronym: GOCol
Status: Completed | Type: Observational
Sponsor: University of Pisa (Other)
Responsible Party: Principal Investigator, Marinò Michele, Ricercatore (Assistant Professor), University of Pisa
Other Study IDs: GOCol
Record Dates: First submitted 2016-03-17; First posted 2016-03-29 (Estimated); Last update posted 2017-08-14 (Actual); Status verified 2017-08

CONDITIONS: Graves' Ophthalmopathy; Hypercholesterolemia
MeSH Terms: conditions — Graves Ophthalmopathy; Hypercholesterolemia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Graves' Disease: Patients with Graves' disease, without Graves' Orbitopathy
  Interventions: Other: No intervention
- Graves' Orbitopathy: Patients with Graves' disease, with Graves' Orbitopathy
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
The investigators have recently observed retrospectively that the occurrence of Graves' Orbitopathy in patients with Graves' disease is less frequent in patients with normal cholesterol levels, in line with another recent observation suggesting that statins play a protective role in Graves' patients from developing Graves' Orbitopathy. The present study is designed in order to investigate the possible association between Graves' Orbitopathy and high cholesterol level as well as the relation between Graves' Orbitopathy degree and high cholesterol level

ELIGIBILITY:
Inclusion Criteria:

1. Graves' disease with Graves' Orbitopathy
2. Graves' disease without Graves' Orbitopathy

Exclusion Criteria:

1. Previous treatment with radioiodine
2. Previous treatment with thyroidectomy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with Graves' disease, with or without Graves' Orbitopathy, off methimazole since two days to perform radioiodine treatment
Sampling Method: Probability Sample
Enrollment: 250 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Relationship between LDL cholesterol levels and Graves' Orbitopathy | Baseline
  Relationship between the levels of LDL cholesterol and the presence of Graves' Orbitopathy

SECONDARY OUTCOMES:
Relationship between LDL cholesterol levels and the activity of Graves' Orbitopathy | Baseline
  Relationship between the levels of LDL cholesterol and the Graves' Orbitopathy clinical activity score
Relationship between LDL cholesterol levels and the severity of Graves' Orbitopathy | Baseline
  Relationship between the levels of LDL cholesterol the Graves' Orbitopathy severity score (NOSPECS score)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Cisanello-Endocrinology I and II, Pisa, Italy

IPD SHARING:
Plan to Share IPD: No